CLINICAL TRIAL: NCT03594695
Title: Hs-CRP and NLR as Markers of Perioperative Stress in Maternal And Fetal Blood in Different Anesthesia Techniques
Brief Title: Hs-CRP and NLR as Markers of Perioperative Stress
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Hakan Yılmaz, Assoc Prof, Ufuk University
Other Study IDs: hsCRP
Record Dates: First submitted 2018-01-15; First posted 2018-07-20 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Cesarean Delivery Affecting Newborn; Anesthesia; Inflammatory Response
Keywords: cesarean section, anesthesia, hs-CRP, NLR

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group G: Patients undergoing general anesthesia HSCRP and NLR measurement
  Interventions: Diagnostic Test: HSCRP and NLR
- Group R: Patients undergoing spinal anesthesia HSCRP and NLR measurement
  Interventions: Diagnostic Test: HSCRP and NLR

INTERVENTIONS:
Diagnostic Test: HSCRP and NLR — hs-CRP levels and NLR values will be studied from routine blood samples.

SUMMARY:
The stress response to surgery is a result of tissue injury with local and systemic inflammation that contributes to the postoperative outcome. Anesthesia is known to effect perioperative stress response Regional anesthesia modifies stress response through afferent blockage whereas general anesthesia affects the stress response via central modulation. High sensitive C-reactive protein and neutrophil to lymphocyte ratio are used for evaluation of inflammation. The aim of this study was to document the value hs-CRP and NLR in perioperative stress response in two different anesthesia methods applied to term pregnant women undergoing elective ceserean section (C/S).

DETAILED DESCRIPTION:
The stress response to surgery is a result of tissue injury with local and systemic inflammation that contributes to the postoperative outcome. Anesthesia is known to effect perioperative stress response. Regional anesthesia modifies stress response through afferent blockage whereas general anesthesia affects the stress response via central modulation. High sensitive C-reactive protein and neutrophil to lymphocyte ratio are used for evaluation of inflammation. The degree of systemic inflammation has been determined by numerous pro- and anti-inflammatory cytokines.The cytokines control the release of C -reactive protein (CRP) which is an acute phase reactant produced by the liver. CRP is a widely used marker of inflammation and tissue damage. High sensitive C -reactive protein (hs-CRP), is a more sensitive assay for detection of inflammation measured by particle-enhanced immunonephelometry . A rapid increase in hs-CRP may indicate inflammation and tissue damage . Another well-known indicator of inflammation is neutrophil-to-lymphocyte ratio (NLR). NLR correlates strongly with elevated plasma levels of circulating proinflammatory cytokineS. The aim of this study was to document the value hs-CRP and NLR in perioperative stress response in two different anesthesia methods applied to term pregnant women undergoing elective ceserean section (C/S).

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women without chronic diseases at term (36-41 weeks of pregnancy)

Exclusion Criteria:

* refusal to participate,
* chronic diseases (diabetes mellitus, hypertension, heart disease, renal disease, hypo/hyperthyroidism)
* any infections,
* smoking
* contraindications for central neuraxial anesthesia.
* Pregnancies complicated with rupture of membranes, placenta previa, eclampsia/preeclampsia, and abruptio placenta
* fetal anomalies,
* abnormality detected at fetal well-being tests

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This observational study is conducted in cesarean sections
Study Population: The study population is composed of healthy pregnant women without chronic diseases at term (36-41 weeks of pregnancy).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in HSCRP levels | preoperative, postoperative 2nd and 4th hours, fetal cord blood sample (following delivery)
  Measurement of high sensitive C reactive protein levels in different time points in order to evaluate the change in HSCRP levels
Evaluation of the change in NLR | preoperative, postoperative 2nd and 4th hours, fetal cord blood sample (following delivery)
  Measurement of the Neutrophil to Lymphocyte Ratio in different time points in order to evaluate the change in the Neutrophil to Lymphocyte Ratios

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Yılmaz, MD, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Ankara, Balgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Jiang S, Wu Y. Effect of 2 different anesthesia methods on stress response in neurosurgical patients with hypertension or normal: A prospective clinical trial. Medicine (Baltimore). 2016 Aug;95(35):e4769. doi: 10.1097/MD.0000000000004769. PMID 27583931
- [Background] Farzadnia M, Ayatollahi H, Hasan-Zade M, Rahimi HR. A comparative study of vascular cell adhesion molecule-1 and high-sensitive C-reactive protein in normal and preeclamptic pregnancies. Interv Med Appl Sci. 2013 Mar;5(1):26-30. doi: 10.1556/IMAS.5.2013.1.5. Epub 2013 Mar 19. PMID 24265885